CLINICAL TRIAL: NCT01508871
Title: Electrical Interactions in Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0126-A
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2011-08

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiomyopathy
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — No intervention

SUMMARY:
This study will evaluate the relationship of markers of cardiac activation and their determinants. The hypothesis is that these markers will be interrelated.

ELIGIBILITY:
Inclusion Criteria:

* ventricular dysfunction

Exclusion Criteria:

* normal ventricular function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventricular dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada